CLINICAL TRIAL: NCT04322994
Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Use in Pediatric Populations: A Randomized Prospective Multi-Site Trial
Brief Title: THRIVE Use in Pediatric Populations- Multi Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Nationwide Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Boston Children's Hospital (Other); UC Davis Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50881
Record Dates: First submitted 2020-03-21; First posted 2020-03-26 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Oxygen Deficiency; Desaturation of Blood; Hypoventilation; Anesthesia; Adverse Effect
MeSH Terms: conditions — Hypoxia; Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): Control subjects will undergo their scheduled procedure and recovery with the usual care. Following recovery from anesthesia, a brief questionnaire will be provided to applicable patients or their parents / guardians / representatives.
- Intervention (Experimental): Treatment subjects will undergo the scheduled procedure, with the difference being that a high-flow nasal cannula will be applied prior to the start of the procedure and removed following the procedure's conclusion. While applied, the cannula will deliver high- flow rate oxygen, air, or a mixture of variable oxygen concentration (21-100%) depending on the surgical conditions and requirements. The rate will be set at 1-4L/kg/min with a maximum of 70L/min. Participants in the treatment arm will then proceed to the recovery area as usual. Following recovery from anesthesia, a brief questionnaire will be provided to applicable patients or their parents / guardians / representatives.
  Intervention: Device: High-flow nasal cannula
  Interventions: Device: Transnasal Humidified Rapid-Insufflation Ventilatory Echange

INTERVENTIONS:
Device: Transnasal Humidified Rapid-Insufflation Ventilatory Echange — The use of high-flow nasal cannula to augment the ability to oxygenate and ventilate a patient under general anesthesia.
  Arms: Intervention

SUMMARY:
THRIVE (Transnasal Humidified Rapid-Insufflation Ventilatory Exchange) refers to the use of high-flow nasal cannula to augment the ability to oxygenate and ventilate a patient under general anesthesia. The use of high-flow nasal cannula oxygen supplementation during anesthesia for surgical procedures has been a recent development in the adult population, with limited data analyzing the pediatric population. This study will determine whether high flow nasal cannula oxygen supplementation during surgical or endoscopic procedures can prevent desaturation events in children under anesthesia and improve the outcomes of that surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients less than 18 years of age undergoing general anesthesia for procedures or surgeries

Exclusion Criteria:

* Pregnancy
* Absence of parent or legal guardian able to provide written consent for study participation
* Anatomical or surgical contraindications (epistaxis, basilar skull fractures or abnormalities, nasal surgery or obstruction, nasal fractures, nasal vascular abnormalities), tracheostomy tube
* Emergent surgery for which application of HFNC might delay surgery or might result in increased aspiration risk.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Massachussetts Eye and Ear Harvard Medical School, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from six pediatric sites (Lucile Packard Children's Hospital, Cincinnati Children's hospital, Lurie Children's Hospital, University of Virginia Children's Hospital, Massachusetts Eye and Ear Infirmary, and Boston Children's Hospital between October 2020 and January 2024. The first participant was enrolled on October 21, 2020 and the last participant was enrolled in January 19, 2024.
Groups:
- Control: Participants undergo their scheduled procedure and recovery with the usual care.
- High-flow Nasal Cannula: Participants undergo their scheduled procedure, and also have a high-flow nasal cannula applied prior to the start of the procedure and removed following the procedure's conclusion.
Period: Overall Study
Arm/Group | Control | High-flow Nasal Cannula
Started | 88 | 87
Completed | 71 | 73
Not Completed | 17 | 14

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | High-flow Nasal Cannula | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (5.2) | 4.7 (5.1) | 5.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 20 | 48
  Male | 43 | 53 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 43 | 87
  Black | 1 | 2 | 3
  Hispanic | 13 | 18 | 31
  Asian | 5 | 2 | 7
  Multirace | 2 | 4 | 6
  Missing | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 73 | 144

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 4% Decrease From Baseline in Oxygen Desaturation Index
Description: Oxygen desaturation index is defined as a 4% decrease in saturation from a 120 second rolling mean for greater than 10 seconds; data were recorded every 2 seconds while the procedure was being performed.
Time Frame: Duration of surgery or procedure, which is generally less than 2 hours
Population: Participants who completed the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High-flow Nasal Cannula
Number analyzed (Participants) | 71 | 73
Participants
  Any event | 18 | 11
  1 event | 13 | 9
  2+ events | 5 | 2
Statistical Analysis 1: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with any desaturation event; Test type: Other; p = 0.18, Chi-squared — The a priori threshold for statistical significance was 0.05; Chi-squared test of independence
Statistical Analysis 2: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with 1 desaturation event versus 2 or more events; Test type: Other; p = 0.26, Chi-squared — The a priori threshold for statistical significance was 0.05; Chi-squared test of independence

2. Primary Outcome: Number of Participants With Desaturations <90%
Description: Relative incidence of oxygen desaturation less than 90% as measured by pulse oximetry by second adjusted for post surgical diagnosis; data were recorded every 2 seconds while the procedure was being performed.
Time Frame: Duration of surgery or procedure, which is generally less than 2 hours
Population: Participants who completed the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High-flow Nasal Cannula
Number analyzed (Participants) | 71 | 73
Participants
  Any event | 17 | 11
  1 event | 8 | 9
  2+ events | 9 | 2
Statistical Analysis 1: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with at any qualifying desaturation event; Test type: Other; p = 0.26, Chi-squared — The a priori threshold for statistical significance was 0.05; Chi-squared test of independence
Statistical Analysis 2: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with 1 qualifying desaturation event versus 2 or more qualifying events; Test type: Other; p = 0.08, Chi-squared — The a priori threshold for statistical significance was 0.05; Chi-squared test of independence

3. Primary Outcome: Number of Participants Who Ever Either Fall Below 90% O2 or Drop 4% Below Baseline Saturation
Description: Relative incidence of oxygen desaturation less than 90% as measured by pulse oximetry by second adjusted for post surgical diagnosis; data were recorded every 2 seconds while the procedure was being performed. Participants who experienced both a fall below 90% O2 and a 4% drop below baseline saturation are reported as having more than 1 event.
Time Frame: Duration of surgery or procedure, which is generally less than 2 hours
Population: Participants who completed the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High-flow Nasal Cannula
Number analyzed (Participants) | 71 | 73
Participants
  Any event | 19 | 13
  1 event | 3 | 3
  2+ events | 16 | 10
Statistical Analysis 1: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with any qualifying event; Test type: Other; p = 0.28, Chi-squared
Statistical Analysis 2: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with 1 qualifying event versus 2 or more events; Test type: Other; p = 0.38, Chi-squared — The a priori threshold for statistical significance was 0.05

4. Secondary Outcome: Time-normalized Area Under Curve (AUC) of Desaturations <90%
Description: Duration of oxygen desaturation less than 90% as measured by pulse oximetry by second by analyzing area under curve less than 90% (in those participants who experienced desaturation less than 90%), normalized as area under the curve / total time.
Time Frame: Duration of surgery or procedure, which is generally less than 2 hours
Population: Participants who experienced desaturation less than 90%
Measure: Mean (Standard Error); unit: % of blood oxygen saturation
Arm/Group | Control | High-flow Nasal Cannula
Number analyzed (Participants) | 17 | 11
% of blood oxygen saturation | 0.3 (0.91) | 0.28 (1.19)
Statistical Analysis 1: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with at any qualifying desaturation event; Test type: Other; p = 0.88, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

5. Secondary Outcome: Number of Participants With Surgical Interruptions Due to Desaturation
Description: Number of surgical interruptions due to desaturation defined by a pause in surgical procedures due to need to provide airway intervention to improve patient's oxygen saturation, normalized to case length. Airway interventions may include jaw thrust, bag mask ventilation, and/or endotracheal intubations.
Time Frame: Duration of surgery or procedure, which is generally less than 2 hours
Population: Participants who completed the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High-flow Nasal Cannula
Number analyzed (Participants) | 71 | 73
Participants
  Any event | 14 | 7
  1 event | 11 | 5
  2+ events | 3 | 2
Statistical Analysis 1: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with any surgical interruption; Test type: Other; p = 0.14, Chi-squared, Corrected — The a priori threshold for statistical significance was 0.05; Chi-squared test of independence
Statistical Analysis 2: Comparison: Control vs High-flow Nasal Cannula; Analysis of between-group difference for participants with 1 surgical interruption versus 2 or more interruptions; Test type: Other; p = 0.21, Chi-squared — The a priori threshold for statistical significance was 0.05; Chi-squared test of independence

6. Secondary Outcome: Minimum Oxygen Saturation as a Measure of Desaturation Severity
Description: Number of participants categorized by lowest oxygen saturation level during surgery (nadir). Lower saturation levels correspond to a lower level of oxygen in red blood cells.
Time Frame: Duration of surgery or procedure by second, which is generally less than 2 hours
Population: Participants who completed the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | High-flow Nasal Cannula
Number analyzed (Participants) | 71 | 73
Participants
  0-50% O2 saturation | 2 | 2
  50-70% O2 saturation | 3 | 2
  70-90% O2 saturation | 12 | 7
  90-100% O2 saturation | 54 | 62

7. Other Pre Specified Outcome: Gas Pain or Bloating
Description: Incidence of gas pain or bloating as measured by post-operative survey
Time Frame: Evaluated postoperatively in post-anesthesia recovery unit prior to discharge, which is about 60 minutes postoperatively
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Nasal Irritation
Description: Incidence of nasal irritation as measured by post-operative survey
Time Frame: as for outcome 7
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Sinus Pressure / Pain
Description: Incidence of sinus pressure and/or pain as measured by post-operative survey
Time Frame: as for outcome 7
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Headache
Description: Incidence of headache as measured by post-operative survey
Time Frame: as for outcome 7
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Other Adverse Events
Description: Other adverse events as measured by post-operative survey
Time Frame: as for outcome 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 days
Arm/Group | Control | High-flow Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/87
Other Adverse Events (participants affected / at risk) | 0/88 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04322994/Prot_SAP_000.pdf